CLINICAL TRIAL: NCT04006548
Title: To Explore the Influence of Appetite Reduction and Medication Effect of Methylphenidate in Patients With Attention-deficit/Hyperactivity Disorder Through Pharmacogenetics.
Brief Title: To Explore the Influence of Appetite Reduction and Medication Effect of Methylphenidate in Patients With Attention-deficit/Hyperactivity Disorder(ADHD) Through Pharmacogenetics.
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CGMH-IRB-201900009B0
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Methylphenidate Adverse Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We plan to recruit 200 children and adolescents aged between 6 to 17 years old in two years. Those patients would receive clinical interview by child psychiatrists to diagnose as ADHD and to exclude mental retardation, major psychiatric disorders and medical disorders. Moreover, we excluded children who ever received ADHD medication treatment more than one year, or received medication in recent 30 days. Initial assessment includes collecting saliva sample, and complete questionnaires (SNAP-IV), clinical rating (CGI-S) and psychological test (CPT-II, WISC-IV, CANTAB). After 1 month methylphenidate treatment, we would evaluate SNAP-IV, CGI-S, CGI-I and Barkley Psychostimulants Side Effects Rating Scale. We also would collect saliva samples to perform appetite related gene phenotyping to see the association between medication side effect and polymorphism of appetite related genes.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 6 years old to17 years old
* Diagnosis of ADHD.

Exclusion Criteria:

* mental retardation.
* major psychiatric disorders
* major medical disorders.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents aged between 6 to 17 years old, diagnosed as ADHD, and recieved methylphenidate treatment.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Barkley psychostimulants side effect scale | One month methylphenidate use
  This scale included 17 most common side-effects of methylphenidate. The occurrence of each side-effect was rated on a Likert scale ranging from 0 (not a problem) to 9 (severe).
Clinical Global Impression scale-Improvement (CGI-I) | One month methylphenidate use
  This scale was used to evaluate the improvement after medication treatment. It's a Likert scale range from 1 (very much improved) through to 7 (very much worse).

CONTACTS AND LOCATIONS:
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan